CLINICAL TRIAL: NCT00014079
Title: Clinical Significance of Genetic Markers in Colon Cancer
Brief Title: Genetic Markers in Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-934655; CDR0000065549 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: DNA is examined for unstable elements (microsatellite instability and loss of heterozygosity) by analyzing at least 10 separate (CA)n-repeats localized to 5 separate chromosomes (5q, 8p, 15, 17p, and 18q). Loss of heterozygosity is analyzed for at least four chromosomal arms (5q, 8p, 17p, and 18q) and later other chromosomes (e.g., 1, 14, and 22). Immunohistochemistry is used to test for the presence or absence of the genes involved in DNA mismatch repair (hMLH1 and hMSH2).
  Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.
  Interventions: Genetic: DNA stability analysis; Genetic: loss of heterozygosity analysis; Genetic: microsatellite instability analysis

INTERVENTIONS:
Genetic: DNA stability analysis
Genetic: loss of heterozygosity analysis
Genetic: microsatellite instability analysis

SUMMARY:
RATIONALE: Determination of genetic markers for colorectal cancer may improve the identification of patients who are at highest risk for relapse.

PURPOSE: This clinical trial is studying the importance of genetic markers for detecting relapse in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical and pathologic significance of unstable DNA elements in colorectal cancer (tumor microsatellite instability).
* Determine the clinical and pathologic significance of loss of heterozygosity for chromosomes 5, 8, 17, and 18 (as the primary targets) and of chromosomes 1, 14, and 22 (as the secondary targets) in colorectal cancer.

OUTLINE: DNA is examined for unstable elements (microsatellite instability and loss of heterozygosity) by analyzing at least 10 separate (CA)n-repeats localized to 5 separate chromosomes (5q, 8p, 15, 17p, and 18q). Loss of heterozygosity is analyzed for at least four chromosomal arms (5q, 8p, 17p, and 18q) and later other chromosomes (e.g., 1, 14, and 22). Immunohistochemistry is used to test for the presence or absence of the genes involved in DNA mismatch repair (hMLH1 and hMSH2).

Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: This study will accrue up to 708 specimens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have had a resectable adenocarcinoma of the colon or rectum and must have participated in one of the following NCCTG randomized clinical trials:

  * 784852: No Treatment Control Versus Levamisole Versus Levamisole Plus Fluorouracil (5-FU)
  * 794604: No Treatment Control Versus 5-FU by Portal Vein Infusion
  * 794751: Postoperative Radiation Versus Postoperative Radiation Plus Sequential Chemotherapy with Methyl CCNU and 5-FU
  * 844652: An Intergroup Study - An Evaluation of Levamisole Plus 5-FU as Surgical Adjuvant Treatment for Resectable Adenocarcinoma of the Colon
  * 864751: Phase III Protocol for Surgical Adjuvant Therapy of Rectal Carcinoma: A Controller Evaluation of (A) Protracted-Infusion 5-FU as a Radiation Enhancer and (B) 5-FU Plus Methyl-CCNU Chemotherapy
  * 874651: M/N - A Controller Evaluation of Recombinant Interferon-gamma (IFL GM) and 5-FU and Folinic Acid With or Without Levamisole as Adjuvant Treatment for Resectable Adenocarcinoma of the Colon
  * 894651: A Controller Phase III Evaluation of 5-FU Combined With Levamisole and Leucovorin as Adjuvant Treatment for Resectable Colon Cancer
* Tissue blocks from the primary colorectal cancer must have been received by the NCCTG operations office

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients have resectable adenocarcinoma of the colon or rectum and has been previously enrolled on N784852, N794604, N844652, N864751, N874651, and N894651.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 1997-09; Primary Completion 2003-07 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Determine the clinical and pathologic significance of unstable DNA elements | Up to 5 years

SECONDARY OUTCOMES:
Determine the clinical and pathologic significance of loss of heterozygosity | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Ribic CM, Sargent DJ, Moore MJ, Thibodeau SN, French AJ, Goldberg RM, Hamilton SR, Laurent-Puig P, Gryfe R, Shepherd LE, Tu D, Redston M, Gallinger S. Tumor microsatellite-instability status as a predictor of benefit from fluorouracil-based adjuvant chemotherapy for colon cancer. N Engl J Med. 2003 Jul 17;349(3):247-57. doi: 10.1056/NEJMoa022289. PMID 12867608